CLINICAL TRIAL: NCT02612246
Title: Randomized, Double-blind, Placebo-controlled, Dose-escalation Study for the Assessment of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of GLPG1972 in Healthy Male Subjects
Brief Title: First-in-Human Single and Multiple Dose of GLPG1972
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1972-CL-101; 2015-004156-21 (EudraCT Number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLPG1972 single dose (Experimental): Single oral dose of GLPG1972 solution - ascending doses
  Interventions: Drug: GLPG1972 single ascending doses
- Placebo single dose (Placebo Comparator): Single oral dose of placebo solution
  Interventions: Drug: Placebo single dose
- GLPG1972 multiple doses (Experimental): Multiple oral doses of GLPG1972 solution - ascending doses
  Interventions: Drug: GLPG1972 multiple ascending doses
- Placebo multiple doses (Placebo Comparator): Multiple oral doses of placebo solution
  Interventions: Drug: Placebo multiple doses

INTERVENTIONS:
Drug: GLPG1972 single ascending doses — single dose, oral solution
  Arms: GLPG1972 single dose
Drug: Placebo single dose — single dose, oral solution, matching placebo
  Arms: Placebo single dose
Drug: GLPG1972 multiple ascending doses — multiple doses, daily for 14 days, oral solution
  Arms: GLPG1972 multiple doses
Drug: Placebo multiple doses — multiple doses, daily for 14 days, oral solution
  Arms: Placebo multiple doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of GLPG1972 given to healthy subjects, compared to placebo. Also, the safety and tolerability of multiple ascending oral doses of GLPG1972 given to healthy subjects daily for 14 days compared to placebo, will be evaluated.

Furthermore, during the course of the study after single and multiple oral dose administrations, the amount of GLPG1972 present in the blood and urine (pharmacokinetics) will be characterized.

The effect of food on the pharmacokinetics of GLPG1972 will also be evaluated. The potential of cytochrome P450 (CYP)3A4 interaction after repeated dosing with GLPG1972 will be explored as well.

During the course of the study after multiple oral dose administrations, the effect of GLPG1972 on biomarkers present in the blood (pharmacodynamics) will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-50 years of age
* Subjects must have a body mass index between 18-30 kg/m²
* Subjects must be judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram and laboratory profile

Exclusion Criteria:

* A subject with a known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device investigational research study
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* Current sexually active (and/or child wish) male; a contraception method should be used

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in number of subjects with adverse events | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1972 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of adverse events
Change versus placebo in number of subjects with abnormal laboratory parameters | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1972 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal laboratory parameters
Change versus placebo in number of subjects with abnormal vital signs | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1972 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal vital signs
Change versus placebo in number of subjects with abnormal electrocardiogram | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1972 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal electrocardiograms
Change versus placebo in number of subjects with abnormal physical examination | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1972 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal physical examination

SECONDARY OUTCOMES:
The amount of GLPG1972 in plasma | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of GLPG1972 in plasma over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects, fasted or fed
The amount of GLPG1972 in urine | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of GLPG1972 in urine over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects, fasted or fed
Ratio of 6-b-hydroxycortisol/cortisol in urine | Twelve hours before dosing on Day 1 and Day 14
  To assess the potential of CYP3A4 interaction after repeated oral dosing with GLPG1972 by means of the ratio of 6-b-hydroxycortisol/cortisol in urine
Levels of GLPG1972 biomarker in blood | Between Day 1 predose and 48 hours after the last dose
  To assess the pharmacodynamics (PD) of GLPG1972 by means of reduction of levels of biomarker in blood by GLPG1972 compared to placebo after repeated oral dosing

CONTACTS AND LOCATIONS:
Overall Officials: Ennis Lee, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium